CLINICAL TRIAL: NCT02613325
Title: Pilot Study to Determine the Feasibility and Functionality of fPAM Imaging for the in Vivo Depth Measurement of Pigmented Lesions and Melanoma Depth
Brief Title: fPAM for the in Vivo Depth Measurement of Pigmented Lesions and Melanoma Depth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201410125
Record Dates: First submitted 2015-11-12; First posted 2015-11-24 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Pigmented Skin Lesion; Melanoma
Keywords: Melanoma; Imaging; Pigmented Lesions; Melanoma Management
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1: fPAM imaging & Single cell PAM imaging (Experimental): * fPAM imaging will be performed prior to scheduled excision. The time to excision will not be extended longer than 2 weeks for imaging purposes.
  * When the participant presents for imaging, the area of the thickest lesion depth will be determined by fPAM. The area of deepest thickness will be marked perpendicular to the longest axis of the lesions and a clinical photo will be taken and placed in the image storage database.
  * Surgical excision will be performed as standard of care and fPAM depth will be compared with histological examination.
  * To image CTCs in cutaneous blood vessels, a small cuticle area on a finger will be imaged (Single cell PAM imaging) and the most distal cutaneous metastasis or metastasis of largest diameter will be imaged
  Interventions: Device: Functional photoacoustic microscopy; Procedure: Standard of care surgical excision; Device: Single cell photoacoustic microscopy

INTERVENTIONS:
Device: Functional photoacoustic microscopy — -Hybrid imaging technique that detects absorbed diffusive protons ultrasonically through the photoacoustic effect.
  Other Names: fPAM
Procedure: Standard of care surgical excision
Device: Single cell photoacoustic microscopy
  Other Names: Single cell PAM

SUMMARY:
The investigators propose the use of functional photoacoustic microscopy (fPAM) to evaluate both benign and malignant pigmented lesions for tumor depth. Through fPAM analysis followed by histological examination, the investigators anticipate that they will be able to non-invasively determine tumor depth of pigmented lesions (moles and melanoma). In melanoma, tumor depth (Breslow's depth) is not only an important prognostic indicator, but also directs surgical treatment. The ultimate goal is to develop a sensitive clinical tool that will allow non-surgical evaluation of pigmented lesions, which eventually, will aid in melanoma diagnosis and management - potentially an earlier and more definitive surgical management.

In addition, the investigators propose to use the combination of fPAM and single-cell PAM to respectively image CTCs in trunk vessels and cuticle capillaries. Based on the investigators' murine models, the investigators anticipate that they will be able to differentiate CTCs from other blood cells and reliably calculate CTC concentration in a non-invasive manner. CTC concentration has been demonstrated to be a valuable indicator of a melanoma's metastatic potential and a potential tool in evaluating treatment efficacy. The ultimate goal is to develop a sensitive imaging device that will allow accurate evaluation of the risk of melanoma recurrence and metastases, that may facilitate treatment monitoring.

ELIGIBILITY:
Inclusion Criteria:

Outcome Measure #1 and #2

* Healthy individuals with pigmented lesions or a partially biopsied melanoma whose treatment plan includes excision
* Participants must be 18 years or older
* Participants must be able to understand and willing to sign a written informed consent document

Outcome Measures #3 and #4

* Patients with either cutaneous, visceral or brain melanoma metastases.
* Participants must be 18 years or older.
* Participants must be Eastern Cooperative Oncology Group (ECOG) status 0-3.
* Participants must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Minors, pregnant patients, incarcerated individuals, and individuals unable to give informed consent will be excluded from this study
* ECOG status > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
In vivo studies using fPAM pigmented lesions imaging to measure tumor depth | Up to 2 weeks
Validate the lesion depth estimated by fPAM | Up to 2 weeks
  -The thickness as measured by fPAM will be compared with the thickness of the formalin fixed excised lesion.

SECONDARY OUTCOMES:
Feasibility and functionality of fPAM as measured by CTC detection | Up to 2 weeks
Feasibility and functionality of single-cell PAM as measured by CTC detection | Up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Cornelius, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu